CLINICAL TRIAL: NCT01416311
Title: Drug Use Investigation for REVOLADE (Chronic Idiopathic Thrombocytopenic Purpura)
Brief Title: Drug Use Investigation for REVOLADE (ITP)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: 114877; CETB115B1401 (Other: Novartis)
Record Dates: First submitted 2011-06-09; First posted 2011-08-15 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
MeSH Terms: conditions — Purpura | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects prescribed REVOLADE: Subjects with chronic idiopathic thrombocytopenic purpura prescribed REVOLADE during study period
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag

SUMMARY:
To investigate safety and efficacy in the actual use of REVOLADE collected from all subjects receiving the drug until data from a specified number of subjects are accumulated to identify factors considered to influence its safety and efficacy.

<Priority investigation item> Thromboembolism

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic idiopathic thrombocytopenic purpura

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Japanese subjects with chronic idiopathic thrombocytopenic purpura who recieve REVOLADE
Sampling Method: Probability Sample
Enrollment: 5797 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
The number of subjects with any adverse events treated with REVOLADE | 1 year

SECONDARY OUTCOMES:
Appearance of thromboembolism | 1 year
  If thromboembolism is appeared or not in subjects who received REVOLADE will be investigated throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals